CLINICAL TRIAL: NCT03986034
Title: Early Clonal Dynamics During Venetoclax Treatment for Chronic Lymphocytic Leukemia (CLL)
Brief Title: Early Clonal Dynamics During Venetoclax Treatment for Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 190111; 19-H-0111
Record Dates: First submitted 2019-06-13; First posted 2019-06-14 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12-15

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: ramp-up; Rituximab; Tumor; Treatment; Cancer
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relapsed/Refractory CLL pts (Experimental): Ages 18 and older
  Interventions: Drug: During Venetoclax

INTERVENTIONS:
Drug: During Venetoclax — Patients with CLL/SLL will enroll on the study. Subjects will be treated at the NIH Clinical Center for the duration of the ramp-up phase of venetoclax. After the ramp-up phase is complete, subjects will be transitioned to the care of their local hematologist/oncologist and receive venetoclax monotherapy or in combination with other agent(s) at the discretion of the treating oncologist. Subjects will have the option to follow-up at the NIH every 6 months (from initiation of venetoclax) and at (suspected) progression.

SUMMARY:
Background:

The drug venetoclax treats chronic lymphocytic leukemia (CLL). Researchers want to find better treatments for CLL. To do that, they need to learn how the drug affects CLL cancer cells and the immune system.

Objective:

To learn about genetic changes that happen during treatment of CLL with venetoclax.

Eligibility:

Adults ages 18 and older with relapsed or refractory CLL after at least 1 prior therapy

Design:

Participants will be screened under a separate protocol.

In Phase 1, participants will get venetoclax free of charge through the NIH. Venetoclax is started at a low dose. The dose will be increased every week until participants reach their maximum tolerable dose. This usually take about 5 weeks. Participants will visit the NIH at least once per week. Visits will be about 4 hours. They may have to stay in the hospital to be observed.

In Phase 2, participants will continue to get the drug through their local cancer doctor and their health insurance. Patients will also visit the NIH every 6 months, or if their disease progresses.

At the NIH participants will have regular health assessments. These will include physical exams and a review of the medicines they are taking. They will talk about how they are feeling.

The study included the following tests:

Blood draws

CT scans: Participants will lie in a machine that takes pictures of the body (maximum 3 per year)

Bone marrow biopsies: A small amount of marrow will be taken out of the participant s hip bone with a needle.

Optional lymph node biopsies: A small piece of the participant s tissue will be taken out with a needle.

The study will last at least 2 years.

DETAILED DESCRIPTION:
This study aims to study the clonal dynamics and kinetics of response during the ramp-up phase of venetoclax in chronic lymphocytic leukemia (CLL).

Key Eligibility Criteria:

1. Diagnosis of CLL/SLL (treatment naive or relapsed/refractory)
2. Must have designated hematologist/oncologist who has agreed to assume care and continue venetoclax after the ramp-up phase is complete
3. Age >=18 years
4. ECOG 0-2

Design:

Patients with CLL/SLL will enroll on the study. Subjects will be treated at the NIH Clinical Center for the duration of the ramp-up phase of venetoclax. After the ramp-up phase is complete, subjects will be transitioned to the care of their local hematologist/oncologist and receive venetoclax monotherapy or in combination with other agent(s) at the discretion of the treating oncologist. Subjects will have the option to follow-up at the NIH every 6 months (from initiation of venetoclax) and at (suspected) progression.

Study Objectives:

Primary Objective:

-Determine the proportion of subjects with clonal shift during the ramp-up phase of venetoclax

Secondary Objective:

-Determine response kinetics of venetoclax therapy in the peripheral blood, lymph nodes and bone marrow

Exploratory Objectives:

* Assess relationship between clonal shifts and minimal residual disease (MRD) status, progression free survival (PFS) and overall survival (OS)
* Assess immunologic changes in the peripheral blood and bone marrow during venetoclax treatment
* Assess circulating-tumor DNA in response to treatment during venetoclax treatment
* Compare the proportion of subjects with early clonal shift between patients receiving only venetoclax and patients receiving venetoclax and BTKi overlap during the ramp-up

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Diagnosis of CLL/SLL which is made according to the updated criteria of the NCI Working Group.
2. Active disease as defined by at least one of the following (iwCLL consensus criteria):

   * Weight loss >=10% within the previous 6 months
   * Extreme fatigue
   * Fevers of greater than 100.5 degrees F for >=2 weeks without evidence of infection
   * Night sweats for more than one month without evidence of infection
   * Evidence of progressive marrow failure as manifested by the development of, or worsening of

     * Anemia and/or thrombocytopenia
     * Massive or progressive splenomegaly
     * Massive nodes or clusters or progressive lymphadenopathy
     * Progressive lymphocytosis with an increase of >50% over a 2-month period, or an anticipated doubling time of less than 6 months
3. Must have designated hematologist/oncologist will assume care and provide venetoclax after the ramp-up phase is complete
4. Must have G6PD testing performed to determine whether rasburicase can be given
5. Must have HLA-testing performed to determine whether allopurinol hypersensitivity exists
6. Age >=18 years
7. ECOG 0-2
8. Agreement to use acceptable methods of contraception for the duration of venetoclax treatment if sexually active and able to bear or beget children
9. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty
10. Able to comprehend the investigational nature of the protocol and provide informed consent

EXCLUSION CRITERIA:

1. Female patients who are currently pregnant or nursing
2. Any uncontrolled active systemic infection
3. Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator s opinion, could compromise the subject s safety or put the study outcomes at undue risk
4. Known additional malignancy that is progressing or requires active treatment.

   --Note: Exceptions include basal cell carcinoma of skin, squamous cell carcinoma of skin, and in situ cervical cancer that has undergone potentially curative therapy. Further exceptions include other cancers from which the subject has been diseasefree for > 2 years, cancers which will not limit survival to < 2 years or cancers in remission receiving endocrine therapy.
5. Richter s Transformation
6. Any prior therapy with BCL-2 inhibitors
7. Concomitant use of strong CYP3A4 inhibitors
8. Disease significantly affecting gastrointestinal function or absorption
9. Uncontrolled autoimmune hemolytic anemia or autoimmune thrombocytopenia
10. Concomitant systemic cancer directed therapy (e.g. immunotherapy, chemotherapy, radiotherapy)
11. Absolute neutrophil count (ANC) <1000/microL, platelets (Plt) <30,000/ microL
12. Serum bilirubin >3 times upper limit of normal (ULN)
13. Severe psychiatric illness/social situations or cognitive impairment that would limit the patient s ability to tolerate and/or comply with study requirements

    * If the PI assesses the decreased ANC and/or Plt to be related to CLL involvement, patients may still be enrolled in the study, as cytopenias as expected to improve with treatment of CLL. Patients may receive supportive measures (e.g. transfusions, IVIG, growth factor support, etc.) to avoid severe cytopenias prior to and during therapy with venetoclax.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-06-26 (Actual); Primary Completion 2026-07-03 (Estimated); Study Completion 2026-07-03 (Estimated)

PRIMARY OUTCOMES:
Determine the rate of clonal shift during the ramp-up phase of venetoclax | 5 weeks.
  The planned analyses will include descriptive statistics on the proportions of clonal shift probability during the venetoclax ramp-up phase. The clonal shift probabilities will be estimated using the sample proportions and their inferences including confidence intervals and hypotheses testing will be evaluated

SECONDARY OUTCOMES:
a. Determine response kinetics of venetoclax therapy in the peripheral blood, lymph nodes and bone marrow | 5 weeks (Primary Endpoint). F/u every 6 months thereafter until disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Gruessner, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
The study team is still deciding.

REFERENCES:
- [Background] Roberts AW, Davids MS, Pagel JM, Kahl BS, Puvvada SD, Gerecitano JF, Kipps TJ, Anderson MA, Brown JR, Gressick L, Wong S, Dunbar M, Zhu M, Desai MB, Cerri E, Heitner Enschede S, Humerickhouse RA, Wierda WG, Seymour JF. Targeting BCL2 with Venetoclax in Relapsed Chronic Lymphocytic Leukemia. N Engl J Med. 2016 Jan 28;374(4):311-22. doi: 10.1056/NEJMoa1513257. Epub 2015 Dec 6. PMID 26639348
- [Background] Herling CD, Abedpour N, Weiss J, Schmitt A, Jachimowicz RD, Merkel O, Cartolano M, Oberbeck S, Mayer P, Berg V, Thomalla D, Kutsch N, Stiefelhagen M, Cramer P, Wendtner CM, Persigehl T, Saleh A, Altmuller J, Nurnberg P, Pallasch C, Achter V, Lang U, Eichhorst B, Castiglione R, Schafer SC, Buttner R, Kreuzer KA, Reinhardt HC, Hallek M, Frenzel LP, Peifer M. Clonal dynamics towards the development of venetoclax resistance in chronic lymphocytic leukemia. Nat Commun. 2018 Feb 20;9(1):727. doi: 10.1038/s41467-018-03170-7. PMID 29463802
- [Background] Stilgenbauer S, Eichhorst B, Schetelig J, Coutre S, Seymour JF, Munir T, Puvvada SD, Wendtner CM, Roberts AW, Jurczak W, Mulligan SP, Bottcher S, Mobasher M, Zhu M, Desai M, Chyla B, Verdugo M, Enschede SH, Cerri E, Humerickhouse R, Gordon G, Hallek M, Wierda WG. Venetoclax in relapsed or refractory chronic lymphocytic leukaemia with 17p deletion: a multicentre, open-label, phase 2 study. Lancet Oncol. 2016 Jun;17(6):768-778. doi: 10.1016/S1470-2045(16)30019-5. Epub 2016 May 10. PMID 27178240
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-H-0111.html